CLINICAL TRIAL: NCT07236489
Title: Prospective Multicenter Randomized Controlled Trial Evaluating the Benefit of Left Bundle Branch Area Stimulation Compared With Conventional Pacing in Post-TAVI Atrioventricular Atrioventricular Block
Brief Title: Trial Evaluating the Benefit of Left Bundle Branch Area Stimulation Compared With Conventional Pacing in Post-TAVI Atrioventricular Atrioventricular Block
Acronym: LBAP-TAVI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC24_0610
Record Dates: First submitted 2025-09-08; First posted 2025-11-19 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Atrioventricular Block; Pacemaker
Keywords: Pacemaker; Atrioventricular block; TAVI; LBAP
MeSH Terms: conditions — Atrioventricular Block

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LBAP : Left Bundle Area Pacing (Experimental): Pacemaker implantation using left bundle branch area stimulation
  Interventions: Procedure: Pacemaker implantation using left bundle branch area stimulation
- RVP : Right Ventricular Pacing (Placebo Comparator): Right ventricular pacemaker implantation
  Interventions: Procedure: Right ventricular pacemaker implantation

INTERVENTIONS:
Procedure: Pacemaker implantation using left bundle branch area stimulation — Pacemaker implantation using left bundle branch area stimulation
  Arms: LBAP : Left Bundle Area Pacing
Procedure: Right ventricular pacemaker implantation — Right ventricular pacemaker implantation
  Arms: RVP : Right Ventricular Pacing

SUMMARY:
Transcatheter aortic valve implantation (TAVI) has rapidly expanded over the past decade as a treatment for severe aortic valve stenosis, with over 14,000 procedures performed in France in 2021. A common complication following TAVI is traumatic atrioventricular block requiring pacemaker implantation, occurring in about 10% of patients. Conventional right ventricular pacing in these cases often leads to interventricular dyssynchrony, which can impair left ventricular ejection fraction and increase the risk of hospitalization, heart failure, and mortality.

Cardiac resynchronization therapy via biventricular pacing is sometimes proposed as a secondary intervention but involves additional surgery. A newer pacing technique-selective left bundle branch area pacing-has been developed to provide physiological ventricular activation by stimulating conduction pathways distal to the lesion, thereby avoiding dyssynchrony. Retrospective studies suggest clinical benefits, but no prospective randomized trial has yet evaluated its efficacy compared to standard pacing.

The objective of this study is to conduct the first randomized clinical trial comparing left bundle branch area pacing versus conventional right ventricular pacing in patients requiring pacemaker implantation due to atrioventricular block after TAVI.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone TAVI for severe aortic valve disease within the past 3 months
* Preserved left ventricular ejection fraction (LVEF ≥ 50%)
* Indications for pacemaker implantation according to guidelines, including :
* Third-degree atrioventricular (AV) block
* Second-degree AV block Mobitz type 2 or symptomatic Mobitz type 1
* Alternating left and right bundle branch block
* HV interval ≥ 70 ms during electrophysiological study
* Pre-existing right bundle branch block with worsening conduction disturbances post-TAVI
* Prolongation of QRS and PR intervals post-procedure justifying pacemaker implantation
* Signed informed consent
* Patient affiliated with the national health insurance system

Exclusion Criteria:

* Left ventricular ejection fraction (LVEF) < 50% before TAVI
* Contraindication to implantation of an endocardial pacemaker (vascular access issues, sepsis)
* Previously implanted pacemaker
* Patients under legal guardianship, curatorship, or judicial protection
* Participation in another interventional therapeutic clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Estimated)
Dates: Start 2025-11-25 (Actual); Primary Completion 2029-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
number of cardiovascular deaths | 24 months
number of hospitalizations for heart failure | 24 months
number of surgical reinterventions | 24 months

SECONDARY OUTCOMES:
success rate of the LBAP technique | 3, 12, and 24 months post-implantation
  Verification of ECG effectiveness criteria: for the LBAP group: qR or rsR' appearance and for the RVP group: QS or rS aspect
comparison of immediate and long-term complications of the LBAP stimulation | 3, 12, and 24 months post-implantation
  Adverse events such as: pneumothorax, infection of equipment, displacement of atrial catheter, lumen haematoma, venous thrombosis, pericardial effusion, reoperation, vascular complication, catheter-specific complications
ECG measurements | 3, 12, and 24 months post-implantation
  QRS duration (ms)
left ventricular function (LVEF) | 3, 12, and 24 months post-implantation
left ventricular diameter | 3, 12, and 24 months post-implantation
creatinine levels | 3, 12, and 24 months post-implantation
GFR in CKD EPI | 3, 12, and 24 months post-implantation
Comparison of the occurrence of atrial fibrillation and ventricular tachycardia (non-sustained or sustained), based on pacemaker monitoring data. | 3, 12, and 24 months post-implantation
EQ-5D-5L questionnaire. | Baseline (inclusion), 3, 12, and 24 months post-treatment
Evaluate the cost-effectiveness of left bundle branch area pacing versus standard therapy in this population using a cost-utility analysis. | 24 months post-implantation
  This will be calculated from EQ-5D-5L utility scores.

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - Brest University Hospital, Brest, Finistère
  - Rennes University Hospital, Rennes, Ille-et-Vilaine
  - Tours University Hospital, Tours, Indre-et-Loire
  - Nantes University Hospital, Nantes, Loire-Atlantique
  - Clermont Ferrand University Hospital, Clermont-Ferrand, Puy-de-Dôme
  - Rouen University Hospital, Rouen, Seine-Maritime
  - Poitiers University Hospital, Poitiers, Vienne